CLINICAL TRIAL: NCT00035438
Title: St. John's Wort Vs. Placebo in Obsessive-Compulsive Disorder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000391-01 (NIH)
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2006-08

CONDITIONS: Obsessive Compulsive Disorder
Keywords: obsessive compulsive disorder; ocd; Anxiety; St. John's Wort; Wisconsin; Psychiatric; Mental health
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Compulsive Personality Disorder; Anxiety Disorders; Psychological Well-Being | interventions — Hypericum extract LI 160

INTERVENTIONS:
Drug: St. John's Wort

SUMMARY:
The purpose of this study is to determine the effectiveness of St. John's Wort as compared to placebo (an inactive substance) in the treatment of outpatients with obsessive compulsive disorder.

DETAILED DESCRIPTION:
The objective of the proposed study is to assess the efficacy of the herbal St. John's Wort (SJW) in the treatment of symptoms of obsessive-compulsive disorder (OCD). The approach is to conduct a 12-week, randomized, double blind, placebo controlled, parallel group pilot trial with 30 subjects in each of two arms. The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) will be the primary measure for evaluating OCD. An intention-to-treat analysis will be done to compare the two arms.

ELIGIBILITY:
Inclusion criteria

* Female patients: at least 2 years post-menopausal, surgically sterile, or practicing a medically acceptable method of contraception.
* Meets DSM-IV criteria for obsessive compulsive disorder

Exclusion criteria

* Primary diagnosis of major depression, dysthymia, panic disorder, social phobia, schizophrenia, schizo-affective disorder, bipolar disorder, or PTSD
* Substance abuse or dependence in the past 6 months
* Vascular dementia or primary degenerative dementia of the Alzheimer's type
* Treatment with MAOIs, TCAs, SSRIs, venlafaxine, nefazodone, remeron, citalopram, or bupropion within 14 days of first visit.
* Fluoxetine within 5 weeks of first visit.
* Failure to respond to at least two adequate antidepressant trials for obsessive compulsive disorder
* Investigational drugs within 30 days of baseline
* Known allergy or hypersensitivity to St. John's Wort
* Currently in behavior therapy for obsessive compulsive disorder

ALL INQUIRIES WILL UNDERGO A PHONE SCREENING TO DETERMINE WHETHER THEY MEET ELIGIBLITY REQUIREMENTS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-05; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kobak, PhD, Principal Investigator — Dean Foundation for Health, Research and Analysis; Leslie Taylo, MD, Principal Investigator — Dean Foundation for Health, Research and Analysis
Locations (2):
- United States (2):
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Dean Foundation, Madison, Wisconsin

REFERENCES:
- See also: A non-profit foundation located in Middleton, Wisconsin, conducting clinical trials of psychiatric and medical therapies. — http://www.dean.org